CLINICAL TRIAL: NCT00624442
Title: A Phase II, Multi Center, Double-Blind, Randomized, Placebo Controlled, Dose-Escalation, Pharmacokinetic (PK) and Pharmacodynamic (PD) Study of CK-1827452 in Patients With Stable Heart Failure
Brief Title: A Study of CK-1827452 Infusion in Stable Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CY 1121
Record Dates: First submitted 2007-12-21; First posted 2008-02-27 (Estimated); Results first posted 2010-08-16 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — omecamtiv mecarbil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (5):
- Cohort 1 (Experimental): 4 treatment periods with a 2 hour infusion. The 4 treatment periods consist of 3 escalating dose levels of CK-1827452 and 1 placebo treatment randomized into the dose escalation sequence. Treatment periods occur at least 7 days apart.
  Interventions: Drug: CK-1827452; Drug: Placebo
- Cohort 2 (Experimental): 4 treatment periods with a 2 hour infusion. The 4 treatment periods consist of 3 escalating dose levels of CK-1827452 and 1 placebo treatment randomized into the dose escalation sequence. Treatment periods occur at least 7 days apart.
  Interventions: Drug: CK-1827452; Drug: Placebo
- Cohort 3 (Experimental): 4 treatment periods with a 24 hour infusion. The 4 treatment periods consist of 3 escalating dose levels of CK-1827452 and 1 placebo treatment randomized into the dose escalation sequence. Treatment periods occur at least 7 days apart.
  Interventions: Drug: Placebo; Drug: CK-1827452
- Cohort 4 (Experimental): 4 treatment periods with a 24 hour infusion. The 4 treatment periods consist of 3 escalating dose levels of CK-1827452 and 1 placebo treatment randomized into the dose escalation sequence. Treatment periods occur at least 7 days apart.
  Interventions: Drug: CK-1827452; Drug: Placebo
- Cohort 5 (Experimental): 2 treatment periods with a 72 hour infusion. The 2 treatment periods are randomly assigned and consist of 1 dose level of CK-1827452 (with dose de-escalation possible depending on tolerability) and 1 placebo treatment. Treatment period 2 occurs at least 7 days after the conclusion of period 1.
  Interventions: Drug: CK-1827452; Drug: Placebo

INTERVENTIONS:
Drug: CK-1827452 — IV infusion for 1 hour at 0.125 mg/kg/h followed by 1 hour at 0.0625 mg/kg/h
  Arms: Cohort 1
Drug: CK-1827452 — IV infusion for 1 hour at 0.25 mg/kg/h followed by 1 hour at 0.125 mg/kg/h
  Arms: Cohort 1
Drug: CK-1827452 — IV infusion for 1 hour at 0.5 mg/kg/h followed by 1 hour at 0.25 mg/kg/h
  Arms: Cohort 1; Cohort 2
Drug: CK-1827452 — IV infusion for 1 hour at 0.75 mg/kg/h followed by 1 hour at 0.375 mg/kg/h
  Arms: Cohort 2
Drug: CK-1827452 — IV infusion for 1 hour at 1.0 mg/kg/h followed by 1 hour at 0.5 mg/kg/h
  Arms: Cohort 2
Drug: CK-1827452 — IV infusion for 1 hour at 0.25 mg/kg/h followed by 1 hour at 0.125 mg/kg/h followed by 22 hours at 0.025 mg/kg/h
  Arms: Cohort 4
Drug: CK-1827452 — IV infusion for 1 hour at 0.5 mg/kg/h followed by 1 hour at 0.25 mg/kg/h followed by 22 hours at 0.05 mg/kg/h
  Arms: Cohort 4
Drug: CK-1827452 — IV infusion for 1 hour at 1.0 mg/kg/h followed by 1 hour at 0.5 mg/kg/h followed by 22 hours at 0.1 mg/kg/h
  Arms: Cohort 4
Drug: Placebo — IV infusion for 2 hours
  Arms: Cohort 1; Cohort 2
Drug: Placebo — IV infusion for 24 hours
  Arms: Cohort 3; Cohort 4
Drug: CK-1827452 — IV infusion for 1 hour at 1.0 mg/kg/h followed 1 hour at 0.5 mg/kg/h followed by 70 hours at 0.1 mg/kg/h
  Arms: Cohort 5
Drug: Placebo — IV infusion for 72 hours
  Arms: Cohort 5
Drug: CK-1827452 — IV infusion for 1 hour at 0.75 mg/kg/h followed 1 hour at 0.5 mg/kg/h followed by 70 hours at 0.1 mg/kg/h
  Arms: Cohort 5
Drug: CK-1827452 — IV infusion for 1 hour at 0.25 mg/kg/h followed by 23 hours at 0.025 mg/kg/h
  Arms: Cohort 3
Drug: CK-1827452 — IV infusion for 1 hour at 0.5 mg/kg/h followed by 23 hours at 0.05 mg/kg/h
  Arms: Cohort 3
Drug: CK-1827452 — IV infusion for 1 hour at 1.0 mg/kg/h followed by 23 hours at 0.1 mg/kg/h
  Arms: Cohort 3

SUMMARY:
This study will assess the safety, tolerability, and pharmacodynamics of CK-1827452 infusion in patients with stable heart failure.

ELIGIBILITY:
Inclusion Criteria

1. Patient is male, or female of non-childbearing potential (two years post-menopausal or surgically sterilized)
2. Female patients must have a negative urine pregnancy test prior to entry into the study
3. Patient is 18 years old or greater
4. Patient has given signed informed consent
5. Patient is considered to be in suitable health in the opinion of the investigator, as determined by:

   * A pre-study physical examination with no clinical abnormalities which in the opinion of the investigator would preclude participation in the study other than physical symptoms or signs consistent with stable heart failure
   * An electrocardiogram (ECG) with no abnormalities in the opinion of the investigator that would impair assessment of stopping criteria
6. Patient has pre-study clinical laboratory findings that are within normal range, or if outside of the normal range, should not preclude participation in the study in the opinion of the investigator (see Exclusion Criteria, below, for exceptions)
7. Patient has a documented diagnosis of heart failure with an ejection fraction of less than 40%
8. Patient has been on a stable dose of a beta blocker and an ACE (angiotensin-converting enzyme) inhibitor or an ARB (angiotensin II receptor blocker) for at least 4 weeks. If prescribed, diuretics must have been administered according to a consistent regimen for at least 4 weeks
9. Patient is currently in sinus rhythm
10. Patient has interpretable echocardiographic images on a screening echocardiogram

Exclusion Criteria

1. Patient has been hospitalized for heart failure, myocardial infarction, coronary revascularization, or another cardiac indication within the last 6 weeks
2. Patient has a current history of alcohol use which in the opinion of the investigator would preclude participation in the study
3. Patient has a current history of drug abuse
4. Patient has donated blood or blood products within 30 days prior to screening
5. Patient has Canadian Cardiovascular Society (CCS) Class III or IV angina
6. Patient has significant obstructive valvular disease or significant congenital heart disease
7. Patient has had a valve replacement
8. Patient is pacemaker dependent
9. Patient is on chronic anti-arrhythmic therapy, with the exception of amiodarone
10. Patient is currently taking, or has taken in the last 7 days, a CYP3A4 inhibitor or inducer medication
11. Patient has a history of hypertrophic obstructive cardiomyopathy
12. Patient weighs > 120 kg
13. Patient has a supine resting systolic blood pressure < 95 mmHg after 3 minutes rest
14. Patient has a supine resting heart rate ≥ 100 beats per minute after 3 minutes rest
15. Patient has an Modification of Diet in Renal Disease (MDRD) estimate of Glomerular Filtration Rate (GFR) ≤ 35 ml/min/1.73 m2
16. Patient has a potassium < 3.5 mEq/L or > 5.5 mEq/L
17. Patient has a sodium ≤ 133 mEq/L
18. Patient has a urea > 15 mmole/L
19. Patient has a troponin I or T at screening that is detectable at the investigative site's clinical laboratory
20. Patient has a hemoglobin < 11 gm/dL in males or < 10 gm/dL in females
21. Patient has an alanine transaminase (ALT), aspartate transaminase (AST), alkaline phosphatase (ALKP) or total bilirubin (TBILI) > 3 times the upper limit of normal
22. Patient is, in the opinion of the investigator, not suitable to participate in the study
23. Patient has participated in any clinical study with an investigational drug within three months prior to the first day of dosing with the exception of coronary stent studies Patient has ever received CK-1827452

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-04; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (2):
  - University of California, San Diego Medical Center, San Diego, California
  - Christiana Care Health Services, Inc., Newark, Delaware
- Diagnostic Services Clinic, Tbilisi, Georgia
- Russia (4):
  - Russian Cardiological Research and Production Complex, Moscow
  - Dzhanelidze Research Institute for Emergency Medical Care, Saint Petersburg
  - Almazov Federal Heart, Blood and Endocrinology Center, Saint Petersburg
  - St. Petersburg State Medical University, Saint Petersburg
- United Kingdom (10):
  - Castle Hill Hospital, University of Hull, Hull, England
  - King's College Hospital, London, England
  - St. George's Hospital, London, England
  - St. Mary's Hospital & Imperial College, London, England
  - Manchester Heart Centre, Manchester Royal Infirmary, Manchester, England
  - ICON Development Solutions, Manchester, England
  - Wythenshawe Hospital, Manchester, England
  - Northwick Park Hospital, Middlesex, England
  - Ninewells Hospital and Medical School, Dundee, Scotland
  - BHF Cardiovascular Centre, Glasgow, Scotland

REFERENCES:
- [Derived] Vu T, Ma P, Xiao JJ, Wang YM, Malik FI, Chow AT. Population pharmacokinetic-pharmacodynamic modeling of omecamtiv mecarbil, a cardiac myosin activator, in healthy volunteers and patients with stable heart failure. J Clin Pharmacol. 2015 Nov;55(11):1236-47. doi: 10.1002/jcph.538. Epub 2015 Jul 14. PMID 25951506
- [Derived] Cleland JG, Teerlink JR, Senior R, Nifontov EM, Mc Murray JJ, Lang CC, Tsyrlin VA, Greenberg BH, Mayet J, Francis DP, Shaburishvili T, Monaghan M, Saltzberg M, Neyses L, Wasserman SM, Lee JH, Saikali KG, Clarke CP, Goldman JH, Wolff AA, Malik FI. The effects of the cardiac myosin activator, omecamtiv mecarbil, on cardiac function in systolic heart failure: a double-blind, placebo-controlled, crossover, dose-ranging phase 2 trial. Lancet. 2011 Aug 20;378(9792):676-83. doi: 10.1016/S0140-6736(11)61126-4. PMID 21856481

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from April 2007 to January 2009.
Groups:
- Cohort 4: 4 treatment periods with a 24 hour infusion. The 4 treatment periods consist of 3 escalating dose levels of CK-1827452 and 1 placebo treatment randomized into the sequence. Treatment periods occur at least 7 days apart.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Started | 8 | 9 | 10 | 8 | 10
Completed | 8 | 8 (One patient was discontinued after inadvertant overdose.) | 8 (Two patients discontinued after meeting termination criteria during dosing.) | 8 | 8 (Two patients discontinued after meeting termination criteria during dosing.)
Not Completed | 0 | 1 | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Total
Number analyzed (Participants) | 8 | 9 | 10 | 8 | 10 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 7 | 6 | 5 | 7 | 30
  >=65 years | 3 | 2 | 4 | 3 | 3 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (11.9) | 56.0 (14.3) | 62.0 (8.2) | 52.6 (18.0) | 57.0 (14.0) | 57.5 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 3 | 2 | 6
  Male | 8 | 8 | 10 | 5 | 8 | 39
Region of Enrollment [Number; unit: participants]
  United States | 0 | 0 | 0 | 1 | 2 | 3
  Georgia | 0 | 0 | 0 | 0 | 2 | 2
  Russian Federation | 0 | 4 | 4 | 2 | 1 | 11
  United Kingdom | 8 | 5 | 6 | 5 | 5 | 29

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Systolic Ejection Time at Various CK-1827452 Plasma Concentrations
Description: Pooled analysis of the echocardiographic measure systolic ejection time from echocardiograms taken at all timepoints. The systolic ejection time is the period during which the aortic valve is open and blood is flowing across the valve. Echocardiograms from cohorts 1,2,3,4 and 5 (564 echocardiograms) were binned into either placebo group or 1 of 6 groups based on plasma concentration of CK-1827452.
Time Frame: 4 days
Population: Pharmacodynamic Population. 4-way crossover design for cohorts 1-4 and 2-way crossover for cohort 5 requires multiple dosing events per participant. Also, multiple PK/PD assessments occur per dosing event.
Measure: Least Squares Mean (Standard Error); unit: msec
Groups:
- >0-100 ng/mL; >100-200 ng/mL; >200-300 ng/mL; >300-400 ng/mL; >400-500 ng/mL; >500 ng/mL: Measurements pooled by plasma concentration of CK-1827452 at time of pharmacodynamic measure. Measurements at any dose level or timepoint could contribute to this bin.
Arm/Group | >0-100 ng/mL | >100-200 ng/mL | >200-300 ng/mL | >300-400 ng/mL | >400-500 ng/mL | >500 ng/mL
Number analyzed (Participants) | 32 | 30 | 27 | 22 | 17 | 25
msec
  # of Echocardiographic Observations (no units) | 84 (0) | 62 (0) | 42 (0) | 24 (0) | 20 (0) | 46 (0)
  Ejection Fraction msec Change from Baseline | 1 (4) | 18 (4) | 47 (5) | 58 (6) | 59 (6) | 80 (5)
Statistical Analysis 1: Comparison: >0-100 ng/mL; Placebo corrected change from baseline least squares mean +/- the standard error of the mean; Test type: Superiority or Other; p = 0.8842, ANCOVA — p-value is not adjusted for multiple comparison Threshold for statistical significance: p<0.05; ANCOVA analysis is based on the following model: CFB Parameter = Bin Group + Baseline + Error, treating patients as a random effect; LSM placebo corrected diff from baseline = 1, 95% CI 2-sided [-7 to 8]
Statistical Analysis 2: Comparison: >100-200 ng/mL; Placebo corrected change from baseline least squares mean +/- the standard error of the mean; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-value is not adjusted for multiple comparison Threshold for statistical significance: p<0.05; [statistical method as in outcome 1, analysis 1]; LSM placebo corrected diff from baseline = 18, 95% CI 2-sided [10 to 27]
Statistical Analysis 3: Comparison: >200-300 ng/mL; Placebo corrected change from baseline least squares mean +/- the standard error of the mean; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-value is not adjusted for multiple comparison Threshold for statistical significance: p<0.05; [statistical method as in outcome 1, analysis 1]; LSM placebo corrected diff from baseline = 47, 95% CI [38 to 56]
Statistical Analysis 4: Comparison: >300-400 ng/mL; Placebo corrected change from baseline least squares mean +/- the standard error of the mean; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-value is not adjusted for multiple comparison Threshold for statistical significance: p<0.05; [statistical method as in outcome 1, analysis 1]; LSM placebo corrected diff from baseline = 58, 95% CI 2-sided [46 to 70]
Statistical Analysis 5: Comparison: >400-500 ng/mL; Placebo corrected change from baseline least squares mean +/- the standard error of the mean; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-value is not adjusted for multiple comparison Threshold for statistical significance: p<0.05; [statistical method as in outcome 1, analysis 1]; LSM placebo corrected diff from baseline = 59, 95% CI 2-sided [47 to 72]
Statistical Analysis 6: Comparison: >500 ng/mL; Placebo corrected change from baseline least squares mean +/- the standard error of the mean; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-value is not adjusted for multiple comparison Threshold for statistical significance: p<0.05; [statistical method as in outcome 1, analysis 1]; LSM placebo corrected diff from baseline = 80, 95% CI 2-sided [71 to 89]
Statistical Analysis 7: Comparison: >0-100 ng/mL vs >100-200 ng/mL vs >200-300 ng/mL vs >300-400 ng/mL vs >400-500 ng/mL vs >500 ng/mL; All available concentration data are used in the model as a continuous variable. p-value based on individual plasma concentration of CK-1827452 vs. corresponding systolic ejection time PD assessment (not binned based on plasma concentration); Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for statistical significance: p<0.05; ANCOVA analysis based on the following model: Change from baseline = Concentration + Baseline + Error, treating patients as random effect

2. Primary Outcome: Change From Baseline of Fractional Shortening at Various CK-1827452 Plasma Concentrations
Description: Pooled analysis of the echocardiographic measure fractional shortening from echocardiograms taken at all timepoints. Fractional shortening is the percentage of change from baseline in the left ventricular cavity dimension with systole. Echocardiograms from cohorts 1,2,3,4 and 5 (564 echocardiograms) were binned into either placebo group or 1 of 6 groups based on plasma concentration of CK-1827452.
Time Frame: 4 days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | >0-100 ng/mL | >100-200 ng/mL | >200-300 ng/mL | >300-400 ng/mL | >400-500 ng/mL | >500 ng/mL
Number analyzed (Participants) | 31 | 28 | 25 | 21 | 14 | 23
Percentage of change
  # of Echocardiographic Observations (no units) | 81 (0) | 56 (0) | 37 (0) | 23 (0) | 17 (0) | 44 (0)
  Fractional Shortening Percent Change from Baseline | 1 (1) | 1 (1) | 3 (1) | 3 (1) | 2 (1) | 5 (1)
Statistical Analysis 1: Comparison: >0-100 ng/mL; Placebo corrected change from baseline least squares mean +/- the standard error of the mean; Test type: Superiority or Other; p = 0.3665, ANCOVA — p-value is not adjusted for multiple comparison Threshold for statistical significance: p<0.05; [statistical method as in outcome 1, analysis 1]; LSM placebo corrected diff from baseline = 1, 95% CI 2-sided [-1 to 2]
Statistical Analysis 2: Comparison: >100-200 ng/mL; Placebo corrected change from baseline least squares mean +/- the standard error of the mean; Test type: Superiority or Other; p < 0.0357, ANCOVA — p-value is not adjusted for multiple comparison Threshold for statistical significance: p<0.05; [statistical method as in outcome 1, analysis 1]; LSM placebo corrected diff from baseline = 1, 95% CI 2-sided [0 to 3]
Statistical Analysis 3: Comparison: >200-300 ng/mL; Placebo corrected change from baseline least squares mean +/- the standard error of the mean; Test type: Superiority or Other; p = 0.0004, ANCOVA — p-value is not adjusted for multiple comparison Threshold for statistical significance: p<0.05; [statistical method as in outcome 1, analysis 1]; LSM placebo corrected diff from baseline = 3, 95% CI 2-sided [1 to 5]
Statistical Analysis 4: Comparison: >300-400 ng/mL; Placebo corrected change from baseline least squares mean +/- the standard error of the mean; Test type: Superiority or Other; p = 0.0086, ANCOVA — p-value is not adjusted for multiple comparison Threshold for statistical significance: p<0.05; [statistical method as in outcome 1, analysis 1]; LSM placebo corrected diff from baseline = 3, 95% CI 2-sided [1 to 4]
Statistical Analysis 5: Comparison: >400-500 ng/mL; Placebo corrected change from baseline least squares mean +/- the standard error of the mean; Test type: Superiority or Other; p = 0.032, ANCOVA — p-value is not adjusted for multiple comparison Threshold for statistical significance: p<0.05; [statistical method as in outcome 1, analysis 1]; LSM placebo corrected diff from baseline = 2, 95% CI 2-sided [0 to 5]
Statistical Analysis 6: Comparison: >500 ng/mL; Placebo corrected change from baseline least squares mean +/- the standard error of the mean; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-value is not adjusted for multiple comparison Threshold for statistical significance: p<0.05; [statistical method as in outcome 1, analysis 1]; LSM placebo corrected diff from baseline = 5, 95% CI 2-sided [3 to 6]
Statistical Analysis 7: Comparison: >0-100 ng/mL vs >100-200 ng/mL vs >200-300 ng/mL vs >300-400 ng/mL vs >400-500 ng/mL vs >500 ng/mL; All available concentration data are used in the model as a continuous variable. p-value based on individual plasma concentration of CK-1827452 vs. corresponding fractional shortening PD assessment (not binned based on plasma concentration); Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for statistical significance: p<0.05; [statistical method as in outcome 1, analysis 7]

3. Secondary Outcome: CK-1827452 Maximum Observed Plasma Concentration (Cmax)
Description: Determined by evaluation of plasma concentrations from blood samples collected prior to dosing and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 12, 24 and 48 hours after initiation of study drug infusion
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: nanogram/milliliter
Groups:
- Cohort 1/2: 0.125 mg/kg/h + 0.0625 mg/kg/h: Subjects received the following CK-1827452 regimen: 0.125 mg/kg/h IV for 1 hour (loading) + 0.0625 mg/kg/h IV for 1 hour (maintenance)
- Cohort 1/2: 0.25 mg/kg/h + 0.125 mg/kg/h: Subjects received the following CK-1827452 regimen: 0.25 mg/kg/h IV for 1 hour (loading) + 0.125 mg/kg/h IV for 1 hour (maintenance)
- Cohort 1/2: 0.5 mg/kg/h + 0.25 mg/kg/h: Subjects received the following CK-1827452 regimen: 0.5 mg/kg/h IV for 1 hour (loading) + 0.25 mg/kg/h IV for 1 hour (maintenance)
- Cohort 1/2: 0.75 mg/kg/h + 0.375 mg/kg/h: Subjects received the following CK-1827452 regimen: 0.75 mg/kg/h IV for 1 hour (loading) + 0.375 mg/kg/h IV for 1 hour (maintenance)
- Cohort 1/2: 1.0 mg/kg/h + 0.5 mg/kg/h: Subjects received the following CK-1827452 regimen: 1.0 mg/kg/h IV for 1 hour (loading) + 0.5 mg/kg/h IV for 1 hour (maintenance)
- Cohort 3: 0.25 mg/kg/h + 0.025 mg/kg/h: Subjects received the following CK-1827452 regimen: 0.25 mg/kg/h IV for 1 hour (loading) + 0.025 mg/kg/h IV for 23 hours (maintenance)
- Cohort 3: 0.5 mg/kg/h + 0.05 mg/kg/h: Subjects received the following CK-1827452 regimen: 0.50 mg/kg/h IV for 1 hour (loading) + 0.05 mg/kg/h IV for 23 hours (maintenance)
- Cohort 3: 1.0 mg/kg/h + 0.1 mg/kg/h: Subjects received the following CK-1827452 regimen: 1.0 mg/kg/h IV for 1 hour (loading) + 0.1 mg/kg/h IV for 23 hours (maintenance)
- Cohort 4: 0.25 mg.kg.h + 0.125 mg/kg/h + 0.025 mg/kg/h: Subjects received the following CK-1827452 regimen: 0.25 mg/kg/h IV for 1 hour + 0.125 mg/kg/h IV for 1 hour + 0.025 mg/kg/h IV for 22 hours
- Cohort 4: 0.5 mg/kg/h + 0.25 mg/kg/h + 0.05 mg/kg/h: Subjects received the following CK-1827452 regimen: 0.5 mg/kg/h IV for 1 hour + 0.25 mg/kg/h IV for 1 hour + 0.05 mg/kg/h IV for 22 hours
- Cohort 4: 1.0 mg/kg/h + 0.5 mg/kg/h + 0.1 mg/kg/h: Subjects received the following CK-1827452 regimen: 1.0 mg/kg/h IV for 1 hour + 0.5 mg/kg/h IV for 1 hour + 0.1 mg/kg/h IV for 22 hours
- Cohort 5: 1.0 mg/kg/h + 0.5 mg/kg/h + 0.1 mg/kg/h: Subjects received the following CK-1827452 regimen: 1.0 mg/kg/h IV for 1 hour + 0.5 mg/kg/h IV for 1 hour + 0.1 mg/kg/h IV for 70 hours
- Cohort 5: 0.75 mg/kg/h + 0.375 mg/kg/h + 0.075 mg/kg/h: Subjects received the following CK-1827452 regimen: 0.75 mg/kg/h IV for 1 hour + 0.375 mg/kg/h IV for 1 hour + 0.075 mg/kg/h IV for 70 hours
Arm/Group | Cohort 1/2: 0.125 mg/kg/h + 0.0625 mg/kg/h | Cohort 1/2: 0.25 mg/kg/h + 0.125 mg/kg/h | Cohort 1/2: 0.5 mg/kg/h + 0.25 mg/kg/h | Cohort 1/2: 0.75 mg/kg/h + 0.375 mg/kg/h | Cohort 1/2: 1.0 mg/kg/h + 0.5 mg/kg/h | Cohort 3: 0.25 mg/kg/h + 0.025 mg/kg/h | Cohort 3: 0.5 mg/kg/h + 0.05 mg/kg/h | Cohort 3: 1.0 mg/kg/h + 0.1 mg/kg/h | Cohort 4: 0.25 mg.kg.h + 0.125 mg/kg/h + 0.025 mg/kg/h | Cohort 4: 0.5 mg/kg/h + 0.25 mg/kg/h + 0.05 mg/kg/h | Cohort 4: 1.0 mg/kg/h + 0.5 mg/kg/h + 0.1 mg/kg/h | Cohort 5: 1.0 mg/kg/h + 0.5 mg/kg/h + 0.1 mg/kg/h | Cohort 5: 0.75 mg/kg/h + 0.375 mg/kg/h + 0.075 mg/kg/h
Number analyzed (Participants) | 8 | 9 | 16 | 9 | 6 | 10 | 9 | 8 | 8 | 9 | 7 | 8 | 2
nanogram/milliliter | 96.1 (27.8) | 195.0 (69.4) | 347.1 (108.6) | 558.1 (156.5) | 635.9 (158.0) | 165.3 (51.4) | 279.9 (55.0) | 633.0 (161.5) | 177.9 (103.4) | 403.3 (226.2) | 681.4 (159.2) | 884.5 (316.2) | 726.9 (62.4)

4. Secondary Outcome: CK-1827452 Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Plasma Concentration (AUClast)
Description: as for outcome 3
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: hour x nanogram/milliliter
Arm/Group | Cohort 1/2: 0.125 mg/kg/h + 0.0625 mg/kg/h | Cohort 1/2: 0.25 mg/kg/h + 0.125 mg/kg/h | Cohort 1/2: 0.5 mg/kg/h + 0.25 mg/kg/h | Cohort 1/2: 0.75 mg/kg/h + 0.375 mg/kg/h | Cohort 1/2: 1.0 mg/kg/h + 0.5 mg/kg/h | Cohort 3: 0.25 mg/kg/h + 0.025 mg/kg/h | Cohort 3: 0.5 mg/kg/h + 0.05 mg/kg/h | Cohort 3: 1.0 mg/kg/h + 0.1 mg/kg/h | Cohort 4: 0.25 mg.kg.h + 0.125 mg/kg/h + 0.025 mg/kg/h | Cohort 4: 0.5 mg/kg/h + 0.25 mg/kg/h + 0.05 mg/kg/h | Cohort 4: 1.0 mg/kg/h + 0.5 mg/kg/h + 0.1 mg/kg/h | Cohort 5: 1.0 mg/kg/h + 0.5 mg/kg/h + 0.1 mg/kg/h | Cohort 5: 0.75 mg/kg/h + 0.375 mg/kg/h + 0.075 mg/kg/h
Number analyzed (Participants) | 8 | 9 | 16 | 9 | 6 | 10 | 9 | 8 | 8 | 9 | 7 | 8 | 2
hour x nanogram/milliliter | 1102.2 (257.6) | 2314.3 (640.9) | 4252.7 (1296.7) | 6060.7 (1741.7) | 8495.7 (3178.3) | 3982.7 (1070.2) | 8120.5 (2268.9) | 18450.7 (4747.8) | 4399.0 (1483.2) | 10624.8 (5168.3) | 19394.3 (4230.6) | 59044.6 (17693.2) | 43605.5 (3551.0)

ADVERSE EVENTS:
Time Frame: 5 weeks
Description: Participants were placed in bins based on their first hour loading dose or placebo. Because multiple dosing events occurred in all cohorts and some loading dose overlap occurs between Cohort 1 and 2 as well as between Cohort 3 and 4, participant numbers in this section do not match the numbers in the participant flow section.
Groups:
- Cohorts 1 and/or 2, Loading Dose of 0.125 mg/kg/hr; Cohorts 1 and/or 2, Loading Dose of 0.25 mg/kg/hr; Cohorts 1 and/or 2, Loading Dose of 0.5 mg/kg/hr; Cohorts 1 and/or 2, Loading Dose of 0.75 mg/kg/hr: Loading dose is the first hour of IV infusion.
- Cohorts 1 and/or 2, Loading Dose of 1.0 mg/kg/hr; Cohorts 3 and 4, Loading Dose of 0.25 mg/kg/hr; Cohorts 3 and 4, Loading Dose of 0.5 mg/kg/hr; Cohorts 3 and 4, Loading Dose of 1.0 mg/kg/hr; Cohort 5, Loading Dose of 0.75 mg/kg/hr; Cohort 5, Loading Dose of 1.0 mg/kg/hr: Loading dose is first hour of IV infusion.
- Cohort 2, Loading Dose of 2.2 mg/kg/hr: Loading dose is first hour of IV infusion. This dose level occurred in 1 patient due to accidental overdose.
Arm/Group | Placebo | Cohorts 1 and/or 2, Loading Dose of 0.125 mg/kg/hr | Cohorts 1 and/or 2, Loading Dose of 0.25 mg/kg/hr | Cohorts 1 and/or 2, Loading Dose of 0.5 mg/kg/hr | Cohorts 1 and/or 2, Loading Dose of 1.0 mg/kg/hr | Cohorts 1 and/or 2, Loading Dose of 0.75 mg/kg/hr | Cohort 2, Loading Dose of 2.2 mg/kg/hr | Cohorts 3 and 4, Loading Dose of 0.25 mg/kg/hr | Cohorts 3 and 4, Loading Dose of 0.5 mg/kg/hr | Cohorts 3 and 4, Loading Dose of 1.0 mg/kg/hr | Cohort 5, Loading Dose of 0.75 mg/kg/hr | Cohort 5, Loading Dose of 1.0 mg/kg/hr
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/8 | 0/9 | 0/16 | 0/6 | 0/8 | 1/1 | 1/18 | 1/18 | 0/16 | 0/2 | 0/8
Other Adverse Events (participants affected / at risk) | 8/41 | 1/8 | 0/9 | 1/16 | 4/6 | 0/8 | 1/1 | 6/18 | 4/18 | 1/16 | 1/2 | 2/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=41) | Cohorts 1 and/or 2, Loading Dose of 0.125 mg/kg/hr (N=8) | Cohorts 1 and/or 2, Loading Dose of 0.25 mg/kg/hr (N=9) | Cohorts 1 and/or 2, Loading Dose of 0.5 mg/kg/hr (N=16) | Cohorts 1 and/or 2, Loading Dose of 1.0 mg/kg/hr (N=6) | Cohorts 1 and/or 2, Loading Dose of 0.75 mg/kg/hr (N=8) | Cohort 2, Loading Dose of 2.2 mg/kg/hr (N=1) | Cohorts 3 and 4, Loading Dose of 0.25 mg/kg/hr (N=18) | Cohorts 3 and 4, Loading Dose of 0.5 mg/kg/hr (N=18) | Cohorts 3 and 4, Loading Dose of 1.0 mg/kg/hr (N=16) | Cohort 5, Loading Dose of 0.75 mg/kg/hr (N=2) | Cohort 5, Loading Dose of 1.0 mg/kg/hr (N=8)
Non ST elevation MI in patient with drug overdose (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septicemia in setting of diabetic foot ulcer (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=41) | Cohorts 1 and/or 2, Loading Dose of 0.125 mg/kg/hr (N=8) | Cohorts 1 and/or 2, Loading Dose of 0.25 mg/kg/hr (N=9) | Cohorts 1 and/or 2, Loading Dose of 0.5 mg/kg/hr (N=16) | Cohorts 1 and/or 2, Loading Dose of 1.0 mg/kg/hr (N=6) | Cohorts 1 and/or 2, Loading Dose of 0.75 mg/kg/hr (N=8) | Cohort 2, Loading Dose of 2.2 mg/kg/hr (N=1) | Cohorts 3 and 4, Loading Dose of 0.25 mg/kg/hr (N=18) | Cohorts 3 and 4, Loading Dose of 0.5 mg/kg/hr (N=18) | Cohorts 3 and 4, Loading Dose of 1.0 mg/kg/hr (N=16) | Cohort 5, Loading Dose of 0.75 mg/kg/hr (N=2) | Cohort 5, Loading Dose of 1.0 mg/kg/hr (N=8)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Other Adverse Event table shows treatment emergent adverse events that occurred in two or more patients. Total for Other Adverse Events is the number of patients affected by an adverse event where an adverse event occurred in two or more patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor intends to publish the results of the trial in collaboration with the Investigators.